CLINICAL TRIAL: NCT01377090
Title: A Multicenter, Prospective Cohort Study Using Nailfold VideoCAPillaroscopy(NVC) and Other Factors to Determine the Risk of Developing Digital Ulceration in Patients With Systemic Sclerosis (SSc)
Brief Title: Digital Ulceration
Acronym: CAP
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-052-521
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Systemic Sclerosis; Digital Ulcers
MeSH Terms: conditions — Scleroderma, Systemic; digital ulcers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SSc DU-history subgroup: Systemic sclerosis patients with history of digital ulcers
- SSc with No-DU-history subgroup: Systemic sclerosis patients with no history of digital ulcers

SUMMARY:
The CAP study is a multicenter, observational, clinical study in patients with systemic sclerosis. The study aims at determining the usefulness of nailfold videocapillaroscopy and patient-specific disease-related factors in predicting the occurrence of digital ulcers within a 6-month observation period. Patients with cutaneous forms of systemic sclerosis (limited or diffuse), with or without history of digital ulceration are eligible. The study will enroll 500 patients at 70 centers.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Signed informed consent prior to enrollment
* Male or female, ≥ 18 years of age
* Diagnosis of systemic sclerosis (SSc) according to the American College of Rheumatology and/or limited cutaneous SSc or diffuse cutaneous SSc according to LeRoy criteria

For patients with no history of digital ulcers (DU) and no DU at enrollment only:

- Enrollment must be within 2 years of the first physician-documented non-Raynaud clinical feature

Exclusion Criteria:

* SSc sine scleroderma (without any skin involvement)
* Patients who underwent stem cell transplantation
* Participation in interventional clinical trials within 3 months prior to enrollment and/or during the study
* Inability to undergo Nailfold Videocapillaroscopy (NVC) assessment (e.g., inability to extend fingers sufficiently)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Systemic Sclerosis with or without a history of digital ulcers (DU)
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Occurence of first new digital ulcer (DU) | 6 months
  Occurrence of the first new digital ulcer (DU) within 6 months

CONTACTS AND LOCATIONS:
Locations (50):
- Austria (4):
  - Medizinische Universität Graz, Graz
  - Universitätsklinik für Innere Medizin Wien, Vienna
  - Sozialmedizinisches Zentrum Süd-Kaiser-Franz-Josef-Spital, Vienna
  - Hanusch Krankenhaus der Gebietskrankenkasse, Vienna
- Belgium (3):
  - Université Libre de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- Revmatologický ústav, Prague, Czechia
- France (7):
  - Centre Hospitalier Universitaire Amiens, Amiens
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - CHRU de Lille, hopital Claude Huriez, Service des maladies du sang, Lille
  - CHU Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Groupe Hospitalier Cochin Saint Vincent de Paul, Paris
  - Hôpital Tenon, Paris
- Germany (9):
  - Asklepios Klinikum Bad Abbach, Bad Abbach
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Berlin
  - Sankt Josef-Hospital, Klinikum der Ruhr-Universität Bochum, Bochum-Gerthe
  - Klinik und Poliklinik für Dermatologie und Venerologie der Universität zu Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Halle (Saale), Halle
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Münster, Münster
- Laiko Hospital, Athens, Greece
- Israel (3):
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
- Italy (6):
  - Universita degli Studi di Brescia, Brescia
  - Azienda Ospedaliera "Pugliese Ciaccio" di Catanzaro, Catanzaro
  - Azienda Ospedale San Martino, Genova
  - Ospedale Santa Ciara, Pisa
  - Policlinico Umberto I, Roma
  - Complesso Integrato Columbus, Roma
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands
- Revmatismesykehuset, Lillehammer, Norway
- Hospital Geral de Santo Antonio, Porto, Portugal
- Spain (4):
  - Hospital Sant Pau, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital de Mostoles, Madrid
  - Hospital Doctor Peset, Valencia
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudoise, Lausanne
  - Kantonspital Sankt Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich
- Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul, Turkey (Türkiye)
- United Kingdom (5):
  - Bath Institute for Rheumatic Diseases, Bath
  - Chapel Allerton Hospital, Leeds
  - Royal Free Hospital, London
  - Hope Hospital, Salford
  - Wrightington Hospital, Wigan